CLINICAL TRIAL: NCT06514456
Title: Italian Validation of the State Urge to be Physically Active- Questionnaire (SUPAQ-I) in Patients With Eating Disorders
Acronym: SUPAQ-I
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 49C402
Record Dates: First submitted 2024-05-30; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Feeding and Eating Disorders
Keywords: Eating Disorders; State Urge to be Physically Active; Anorexia Nervosa; Bulimia Nervosa; Binge Eating Disorder; Questionnaire Language Validation; Urge to move; Physical activity
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Eating disorders (EDs) are severe psychiatric conditions that cause significant health and psychosocial issues, with Anorexia Nervosa (AN) and Bulimia Nervosa (BN) having the highest mortality rates. The COVID-19 pandemic has led to an increase in ED cases, especially among children, with heightened restrictive eating and compulsive exercise. Up to 80% of individuals with AN engage in compulsive exercise, which current treatments fail to adequately address.

The State Urge to be Physically Active Questionnaire (SUPA-Q) is the only validated tool for assessing activity urges in ED patients, covering cognitive, emotional, and behavioral aspects. This study aims to develop and validate an Italian version of the SUPA-Q (SUPAQ-I) in a clinical sample of ED patients.

A mixed-longitudinal study design will be used, with assessments at admission (T0) and discharge (T1) to evaluate the SUPAQ-I's reliability, validity, and sensitivity to change. The sample will include patients aged 16-65 diagnosed with EDs undergoing inpatient rehabilitation. Statistical analyses will include exploratory and confirmatory factor analyses, and internal consistency will be measured using Cronbach's α and McDonald's Ω indices.

Validating the SUPAQ-I will improve the assessment of activity urges in ED patients, enhancing treatment strategies and outcomes.

DETAILED DESCRIPTION:
Eating disorders (EDs) are characterized by a persistent disturbance of eating or eating-related behaviour resulting in altered consumption or absorption of food and leading to both life-threatening somatic complications and psychosocial impairment. Like most psychiatric disorders, EDs underlie pathogenetic mechanisms implying the interaction of neurobiological and genetic factors with the environment. EDs cause over 3000 deaths per year with worsening illness course and increasing chronic cases. For people suffering from EDs, quality of life is reduced and yearly healthcare costs are 48% higher than in the general population. Specifically, Anorexia Nervosa and Bulimia Nervosa report the highest mortality rates among EDs and psychiatric disorders in general. Following the outbreak of Covid-19 pandemic, a concerning increase in both hospital admissions rates and outpatient visits was reported worldwide especially in paediatric populations. Along with this surge in ED cases, changes in symptoms manifestation were also reported, especially in terms of increase in restrictive eating, social media use, comorbid anxiety and depression symptoms and compulsive physical exercise. Food obsession, concerns about body shape and weight contribute to favour ED patients engagement in ritualised behaviours such as counting calories, frequent weighing and problematic physical activity (PA), in terms of frequency, duration and intensity. Notably, up to 80% of individuals with AN engage in voluntary compulsive exercise as a form of weight control. Simultaneously, on a neurobiological basis, starvation appear to heightened the urge to move and restlessness in AN. Current interventions for AN primarily focus on addressing various facets of eating disorders, but treatments exhibit limited efficacy in targeting physical exercise, despite the growing recognition of PA as a pivotal factor reinforcing eating pathology. The heightened restlessness activation in AN might also contribute to the overestimation of body size by enhancing proprioception. Thus far, there are just a few validated instruments to assess acute activity urges in ED patients, with the State Urge to be Physically Active Questionnaire (SUPA-Q), being the only one validated in this clinical population and covering several of the cognitive, emotional and specific behavioural aspects related to activity urges. The SUPA-Q, a 21-item self-report questionnaire, has demonstrated high consistency, reliability, as well as convergent, divergent and factorial validity. Sensitivity to change has also been tested (Cohen's d= 0.48). However, to the best of our knowledge, there has been only one validation study of the SUPA-Q. The objective of this study is to evaluate the psychometric properties of the Italian version of the SUPA-Q, and to test its validity in a clinical sample of patients with EDs.

ELIGIBILITY:
Inclusion criteria:

* age between 16 and 65 years old;
* diagnosis of ED as per DSM 5 or DSM-5 TR
* BMI* range between 13 and 30 kg/m2 (depending on ED main diagnosis)
* for the pediatric population BMI SDS** range is set between -3 and +3 SD from expected BMI for age and sex

Exclusion criteria:

* presence of other pathologies not associated with ED (i.e., neurodegenerative diseases);
* severe psychopathologies other than ED (i.e., schizophrenia)

  * BMI will be calculated using the following formula: weight (kg)/height (m2) **For the pediatric population, BMI SDS will also be calculated to adjust BMI according to growth curve charts for children and adolescents belonging to the Italian population

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of both biological sexes affected by ED who will take part in the multidisciplinary inpatient intensive rehabilitation treatment as offered by the U.O. dei Disturbi del Comportamento Alimentare, San Giuseppe Hospital, Piancavallo (VCO), Italy.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Height | through study completion, an average of 24 months
  height in mt
Weight | through study completion, an average of 24 months
  Weight in kg
BMI | through study completion, an average of 24 months
  body mass index (in kg/m2)
State Urge to be Physically Active Questionnaire Italian Version (SUPAQ-I) | through study completion, an average of 24 months
  State Urge to be Physically Active Questionnaire Italian Version (SUPAQ-I): It consists of a 21-item self-report questionnaire on a 5-point Likert scale (not at all, very little somewhat, quite a bit, a great deal). Items are divided into four scales (burden, emotional aspects, cognitive aspects and motor aspects). The higher the score, the greater the restlessness and the "state" urge to be physically active. Min. score: 0; max. score: 84. A decrease in SUPAQ-I scores means a better outcome.

SECONDARY OUTCOMES:
Eating Disorder Inventory-3 (EDI-3) | through study completion, an average of 24 months
  The questionnaire consists of 91 items evaluated on a six-point Likert scale (always, usually, often, sometimes, rarely, never). The 91 items are divided into twelve primary scales (three scales three refer specifically to the eating disorder: drive for thinness (min 7, max 42), bulimia (min 8, max 48), and body dissatisfaction (min 10, max 60); nine general psychological scales relevant but non-specific for eating disorders: low self-esteem (min 6, max 36), personal alienation (min 7, max 42), interpersonal insecurity (min 7, max 42), interpersonal alienation (min 7, max 42), interoceptive deficits (min 9, max 54), emotional dysregulation (min 8, max 48), perfectionism (min 6, max 36), asceticism (min 7, max 42), and maturity fears (min 8, max 48). The higher the score, the greater the severity of the symptoms. A decrease in EDI-3 scores means a better outcome.
Compulsive Exercise Test (CET) | through study completion, an average of 24 months
  The CET consists of a 24-item self-administered questionnaire evaluated on a 6-point Likert scale from 0 (never true) to 5 (always true). Items are divided into four scales (avoidance, weight control, mood, lack of enjoyment and rigidity). The Italian version of the CET showed acceptable reliability (Cronbach's α coefficients for all the domains > .70). The higher the score, the greater the "trait"-like compulsive physical activity (cut-off is set at 15 points). Min score: 0; max. score: 120. A decrease in CET scores means a better outcome.
Exercise Addiction Inventory - Revised (EAI-R) | through study completion, an average of 24 months
  Exercise Addiction Inventory - Revised : The EAI-R consists of a 6-item self-report questionnaire evaluated on a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). The higher the score the strongest the exercise addiction risk. Min score: 6; max score: 36. A decrease in EAI-R scores means a better outcome.
Barratt Impulsiveness Scale (15 item) (BIS-15) | through study completion, an average of 24 months
  Barratt Impulsiveness Scale (15 item): It consists of a 15-item self-report questionnaire evaluated on a 4-point Likert scale from 1 (rarely/never) to 4 (almost always/always). Items are divided into four scales (pure impulsivity, planning and thinking, lack of attention and concentration impulsive buying). The higher the total score, the greater impulsivity. Min score: 15; max score: 60. This questionnaire will be used to test for divergent validity of the SUPAQ-I.

OTHER OUTCOMES:
Age | through study completion, an average of 24 months
  age in years

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Mendolicchio, M.D., Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy